CLINICAL TRIAL: NCT02667314
Title: Jigsaw Puzzles As Cognitive Enrichment
Brief Title: The Effect of Solving Jigsaw Puzzles on Visuospatial Cognition in Older Adults: Jigsaw Puzzles As Cognitive Enrichment
Acronym: PACE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Ulm (Other)
Collaborators: Ravensburger Spieleverlag GmbH (RSV), Germany (Unknown)
Responsible Party: Principal Investigator, Iris Kolassa, Prof. Dr., University of Ulm
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Klipsy_044_PACE
Record Dates: First submitted 2016-01-20; First posted 2016-01-28 (Estimated); Last update posted 2018-11-30 (Actual); Status verified 2018-11

CONDITIONS: Cognitive Impairment
Keywords: Cognition; Cognitive Aging; Dementia; Neurocognitive Disorders; Cognitive Therapy; Cognitive Reserve; Cognitive Enrichment; Jigsaw Puzzles
MeSH Terms: conditions — Cognitive Dysfunction; Dementia; Neurocognitive Disorders

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Jigsaw Puzzle Group (Experimental): Jigsaw puzzles & Cognitive health counseling
  Interventions: Behavioral: Jigsaw puzzles; Behavioral: Cognitive health counseling
- Cognitive Health Counseling Group (Active Comparator): Cognitive health counseling only
  Interventions: Behavioral: Cognitive health counseling

INTERVENTIONS:
Behavioral: Jigsaw puzzles — Intervention period 1: Participants are asked to solve jigsaw puzzles at home 6 times per week for at least 1 hour over a period of 5 weeks.
  Intervention period 2 (voluntary): Participants receive the possibility to solve jigsaw puzzles free-of-charge at home for a period of at least 3 month before the 1.5-year follow-up.
  Arms: Jigsaw Puzzle Group
Behavioral: Cognitive health counseling — Cognitive health counseling regarding modifiable risk and protective factors of cognitive decline and dementia at baseline, and four telephone calls for expert monitoring (three calls during the 5-week period between pre- and posttest, and one call 12 month later)

SUMMARY:
Meta-analyses indicate beneficial effects of cognitive training and cognitively challenging video games on cognition. However, cognitive effects of solving jigsaw puzzles - a popular, visuospatial cognitive leisure activity - have not been investigated, yet. Thus, the primary aim of this study is to evaluate the effect of solving jigsaw puzzles on visuospatial cognition. As secondary aims, effects on psychological outcomes (self-efficacy, perceived stress, well-being) and visuospatial everyday functioning (instrumental activities of daily living and self-reported cognitive failures in everyday life) are examined.

DETAILED DESCRIPTION:
see References section below for the study protocol article

ELIGIBILITY:
Inclusion Criteria:

* No cognitive impairment (Mini-Mental State Examination ≥ 24)
* Commitment to minimum jigsaw puzzle time (1 hour/day, 6 days/week, 5 weeks)
* Interest in jigsaw puzzles
* Low jigsaw puzzle experience (less than 5 completed puzzles within the last 5 years)

Exclusion Criteria:

* Cognitive impairment (Mini-Mental State Examination < 24)
* Participation in another interventional study
* Self-reported psychiatric, neurologic or other disease, which could affect cognitive change over time
* Self-reported, severe visual impairment or motoric impairment of the upper extremity which significantly affects ability to solve jigsaw puzzles

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2016-02; Primary Completion 2018-02 (Actual); Study Completion 2018-02 (Actual)

PRIMARY OUTCOMES:
Change in global visuospatial cognition from baseline to post intervention and to the 1.5-year follow-up | Baseline and post intervention (after 5 weeks and 1.5 years)
  Averaged score of eight z-standardized visuospatial cognitive ability scores (see secondary outcomes 2 - 9)

SECONDARY OUTCOMES:
Change in visual perception from baseline to post intervention and to the 1.5-year follow-up | Baseline and post intervention (after 5 weeks and 1.5 years)
  Judgment of Line Orientation Test
Change in visuoconstruction from baseline to post intervention and to the 1.5-year follow-up | Baseline and post intervention (after 5 weeks and 1.5 years)
  Copying in Complex Figure Tests; parallel versions for baseline and post-test
Change in mental rotation from baseline to post intervention and to the 1.5-year follow-up | Baseline and post intervention (after 5 weeks and 1.5 years)
  Mental Rotations Test-Letters (2D) and Form A (3D)
Change in visuospatial processing speed from baseline to post intervention and to the 1.5-year follow-up | Baseline and post intervention (after 5 weeks and 1.5 years)
  Trail Making Test A
Change in visuospatial flexibility from baseline to post intervention and to the 1.5-year follow-up | Baseline and post intervention (after 5 weeks and 1.5 years)
  Trail Making Test B
Change in visuospatial working memory from baseline to post intervention and to the 1.5-year follow-up | Baseline and post intervention (after 5 weeks and 1.5 years)
  Block span (Wechsler Memory Scale, German version)
Change in visuospatial reasoning from baseline to post intervention and to the 1.5-year follow-up | Baseline and post intervention (after 5 weeks and 1.5 years)
  Block design (Wechsler Adult Intelligence Scale-III, German version)
Change in visuospatial episodic memory from baseline to post intervention and to the 1.5-year follow-up | Baseline and post intervention (after 5 weeks and 1.5 years)
  Recall in Complex Figure Tests (sum score of immediate and delayed recall); parallel versions for baseline and post-test
Change in psychological health from baseline to post intervention and to the 1.5-year follow-up | Baseline and post intervention (after 5 weeks and 1.5 years)
  Averaged score of three z-standardized psychological health sub-scores (see secondary outcomes 11 - 13)
Change in psychological well-being from baseline to post intervention and to the 1.5-year follow-up | Baseline and post intervention (after 5 weeks and 1.5 years)
  WHO-Five Well-being Index (WHO-5), German version
Change in self-efficacy from baseline to post intervention and to the 1.5-year follow-up | Baseline and post intervention (after 5 weeks and 1.5 years)
  General Self-Efficacy Scale, German version
Change in perceived stress from baseline to post intervention and to the 1.5-year follow-up | Baseline and post intervention (after 5 weeks and 1.5 years)
  Perceived Stress Scale-14, German translation
Change in objective everyday functioning from baseline to post intervention and to the 1.5-year follow-up | Baseline and post intervention (after 5 weeks and 1.5 years)
  TIADL (1-3): Timed instrumental activities of daily living (Task 1-3; sum-score)
Change in self-reported everyday functioning from baseline to post intervention and to the 1.5-year follow-up | Baseline and post intervention (after 5 weeks and 1.5 years)
  CFQ (visuospatial items): Cognitive Failures Questionnaire, sum score of visuo-spatial items; German version
Change in jigsaw puzzle performance from baseline to post intervention and to the 1.5-year follow-up | Baseline and post intervention (after 5 weeks and 1.5 years)
  40-pieces mini puzzle (completed pieces per minute)
Hair cortisol concentration at the 1.5-year follow-up | 1.5-year follow-up
  Hair cortisol will be measured in 1cm segements
Hair dehydroepiandrosteron concentration at the 1.5-year follow-up | 1.5-year follow-up
  Hair dehydroepiandrosteron will be measured in 1cm segements
Hair brain-derived neurotrophic factor concentration at the 1.5-year follow-up | 1.5-year follow-up
  Hair brain-derived neurotrophic factor will be measured in 1cm segements
Neurocognitive disorder | 1.5-year follow-up
  Neurocognitive disorder is a categorical outcome and includes mild and major neurocognitive disorders. Mild neurocognitive disorder (mild cognitive impairment) is defined by subjective cognitive decline (self-report), and an objective cognitive impairments in at least one cognitive abilitiy score (below -1 SD of the norm group), without an essential impairment of daily functioning compared to the premorbid level (self-report). In major neurocognitive decline (dementia), in addition to cognitive decline and impairment, daily functioning is essentially impaired compared to the permorbid level (self-report).

CONTACTS AND LOCATIONS:
Overall Officials: Iris-Tatjana Kolassa, Prof., Principal Investigator — University of Ulm, Germany
Locations (1):
- Clinical and Biological Psychology, University of Ulm, Ulm, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Fissler P, Kuster OC, Loy LS, Laptinskaya D, Rosenfelder MJ, von Arnim CAF, Kolassa IT. Jigsaw Puzzles As Cognitive Enrichment (PACE) - the effect of solving jigsaw puzzles on global visuospatial cognition in adults 50 years of age and older: study protocol for a randomized controlled trial. Trials. 2017 Sep 6;18(1):415. doi: 10.1186/s13063-017-2151-9. PMID 28877756
- [Result] Fissler P, Kuster OC, Laptinskaya D, Loy LS, von Arnim CAF, Kolassa IT. Jigsaw Puzzling Taps Multiple Cognitive Abilities and Is a Potential Protective Factor for Cognitive Aging. Front Aging Neurosci. 2018 Oct 1;10:299. doi: 10.3389/fnagi.2018.00299. eCollection 2018. PMID 30327598
- See also: PACE study protocol article (open access) — http://rdcu.be/vEhX
- See also: PACE results for primary outcome at follow-up I (open access) — https://doi.org/10.3389/fnagi.2018.00299